CLINICAL TRIAL: NCT02002793
Title: Effects of Early Stage Mini-invasive Abdominal Drainage on Complications and Prognosis of SAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Erzhen Chen, Professor, Ruijin Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SAP bundle-abdominal drainage
Record Dates: First submitted 2013-11-11; First posted 2013-12-06 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Pancreatitis
Keywords: pancreatitis; early stage; mini-invasive abdominal drainage
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early stage abdominal drainage (Other): SAP patients who matches one of the following criteria:1．Intravesical pressure≥20cmH2O or 2.CT images:acute peripancreatic liquid collection should have early stage abdominal drainage immediately;
  Interventions: Other: Early stage abdominal drainage
- Late stage abdominal drainage (Other): Despite that it matches one of the cirteria as the study group:1．Intravesical pressure≥20cmH2O or 2．CT images:acute peripancreatic liquid collection, the patients continue acquire prearranged integrative treatment and will not accept early stage abdominal drainage until any of the followings emerge:1.Intra-abdominal apartment syndrome; 2. Pancreatic pseudocyst;3. Pancreatic or peripancreatic necrosis;
  Interventions: Other: Late stage abdominal drainage

INTERVENTIONS:
Other: Early stage abdominal drainage — Ultrasound/CT/GUS guided abdominocentesis and drainage with single-chamber deep venous catheters shoule be implemented and the catheter should be removed when abdominal drainage flow≤100ml in two successive days;
  Arms: Early stage abdominal drainage
Other: Late stage abdominal drainage — Despite that it matches one of the cirteria as the study group:1．Intravesical pressure≥20cmH2O or 2．CT scan:acute peripancreatic liquid collection, the patients continue acquire prearranged integrative treatment and will not accept early stage abdominal drainage until any of the followings emerge:1.Intra-abdominal apartment syndrome; 2. Pancreatic pseudocyst;3. Pancreatic or peripancreatic necrosis;
  Arms: Late stage abdominal drainage

SUMMARY:
This study aims to standardized the process of mini-invasive abdominal draniage of SAP in early stage.To determine the indications and occasion.

DETAILED DESCRIPTION:
Pancreatitis associated ascetic fluids(PAAF) gather with the beginning of SAP and induced IAP(intra-abdominal pressure) increasement.With an excess of 12mmHg ,IAP presents as IAH(intra-abdominal hypertension) and when a ≥20mmHg IAP accompanied with at least one organ's dysfunction it is ACS(abdominal compartment syndrome).Previous recommended theraphy of ACS is laparotomy.However,with inherited advantages such as ease-to-operate and minimal invassiveness, early stage mini-invasive abdominal drainage therapies , for example, percutaneous catheter drainage(PCD) instructed by ultrasound or CT ,have shown a promised future in recent years. It is reported that patients acquired PCD decreased 81% in operation rate compared to those who did not and had lower mortality rate. Whereas, the operation flow of early stage mini-invasive abdominal drainage remains controversial, and whose validity calls for evidence from large-scale clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1.Diagnosis of pancreatitis 2.Onset of abdominal pain within 72h 3.Moderate severe or severe AP according to Atlanta criteria revisited in 2012 4.Intravesical pressure≥20cmH2O 4.CT images:acute peripancreatic liquid collection

-

Exclusion Criteria:

1.Pregnancy 2.Heart function: NYHA >II 3.Pacemaker implantation 4.COPD 5.CKD 6.Pre-existing disease with life expectancy < 3 months 7.CT images:No acute peripancreatic liquid collection 8.Intravesical pressure>25cmH2O 9.At least one organ'S newly emerged dysfunction

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-09 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Rates of ACS in 28 days since outbreaks | 28 days
  Time of first attacks of these situations that have to be surgically interfered in 28 days since onsets: ACS or pancreatic necrosis, abdominal hemorrhage, pancreatic abscess or pancreatic pseudocyst which brings symptoms or complications or increase in size;rates of organs' dysfunction, abdominal infection and reuse of drainage;

SECONDARY OUTCOMES:
Rates of surgical interfere, MODS or death in 6 months since outbreaks | 6 months
  Rates of mortality or organs' dysfunction; rates of complications, including: pancreatic leakage, pancreatic pseudocysts in need of surgical interfere, pancreatic abscess, bile duct stricture and pancreatic insufficiency; times of surgery, hospital stay, time in ICU and hospitalization expense;

CONTACTS AND LOCATIONS:
Overall Officials: erzhen Chen, Professor, Study Director — Emergency intensive care unit of Ruijin Hospital
Locations (1):
- Ruijin, Shanghai, Shanghai Municipality, China